CLINICAL TRIAL: NCT02862795
Title: Human PapillomaVirus (HPV) Anal Infection: Study of Prevalence and Risk Factors Among 1000 Patients Benefiting From a Colonoscopy
Brief Title: Human Papillomavirus Anal Infection
Acronym: PAPILLAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: API/2012/34
Record Dates: First submitted 2016-08-04; First posted 2016-08-11 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-08

CONDITIONS: HPV Infection
Keywords: colonoscopy
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HPV detection in anal canal samples (Other)
  Interventions: Procedure: HPV detection in anal canal samples

INTERVENTIONS:
Procedure: HPV detection in anal canal samples — Additional anal taking during the colonoscopy with cytobrush

SUMMARY:
Human papillomavirus (HPV) are involved in up to 95 % of anal canal neoplastic lesions. Little is known about HPV carriage in anal canal previous to cancer occurrence in the population and pre-neoplastic lesions, and their risk factors. PAPILLAN is a prospective study that aims to study HPV infection (HPV low grade and high grade genotypes) prevalence in anal canal in a population non selected by its HIV status. In that purpose patients are prospectively recruited in a french university hospital gastroenterology unit and anal smears are collected during a colonoscopy with cytobrush.

ELIGIBILITY:
Inclusion Criteria:

* patients > 18 years
* patients undergoing colonoscopy under general anesthesia for any purpose
* signed written consent

Exclusion Criteria:

* age under 18
* Absence of written consent.
* patients incapable of giving consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2012-04; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
anal canal HPV infection | at inclusion (the day of colonoscopy)

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre Hospitalier Régional Universitaire de Besançon, Besançon
  - Centre Hospitalier Intercommunal de la Haute Saône, Vesoul